CLINICAL TRIAL: NCT06955598
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Subcutaneous Injections of SHR-2173 in Patients With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-2173-103
Record Dates: First submitted 2025-04-08; First posted 2025-05-02 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-04

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A: (Experimental): SHR-2173 injection dose 1
  Interventions: Drug: SHR-2173
- Treatment group B: (Experimental): SHR-2173 injection dose 2
  Interventions: Drug: SHR-2173
- Treatment group C: (Experimental): SHR-2173 injection dose 3
  Interventions: Drug: SHR-2173

INTERVENTIONS:
Drug: SHR-2173 — SHR-2173

SUMMARY:
To investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of multiple subcutaneous injections of SHR-2173 in patients with systemic lupus erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years, regardless of gender;
2. Weight ≥45.0 kg at screening;
3. Confirmed SLE diagnosis for ≥12 weeks at screening.

Exclusion Criteria:

1. Pregnant or breastfeeding women, or those with a positive human chorionic gonadotropin (HCG) test.
2. History of alcohol abuse or illegal drug use within one year prior to screening.
3. Blood donation ≥450 mL within 8 weeks prior to screening or plans to donate blood during the study.
4. Current active infection or a history of active tuberculosis
5. Other inflammatory or autoimmune diseases beyond SLE and LN that may interfere with the interpretation of trial results or clinical assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-24 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Adverse events | Week 0~16

SECONDARY OUTCOMES:
Cmax, | Week 0~16
AUC0-t, | Week 0~16
Anti- SHR -2173 antibody (ADA) | Week 0~16

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital affiliated to Shanghai Jiaotong, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided